CLINICAL TRIAL: NCT00896402
Title: Chlorhexidine vs. Betadine in Preventing Colonization of Continuous Femoral Catheters After Total Joint Arthroplasty
Brief Title: Chlorhexidine Versus Betadine in Preventing Colonization of Femoral Nerve Catheters After Total Joint Arthroplasty (TJA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding inadequate
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Joseph Marino M.D., Chief of Anesthesiology, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 1989mdmd
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Infection
Keywords: chloraprep; betadine; colonization; femoral catheter
MeSH Terms: conditions — Infections | interventions — Chlorhexidine; Ethanol; Povidone-Iodine; Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine (Active Comparator): skin antisepsis with chlorhexidine
  Interventions: Drug: Skin antisepsis with chlorhexidine
- Povidone-iodine (Active Comparator): skin antisepsis with povidone-iodine
  Interventions: Drug: povidone-iodine

INTERVENTIONS:
Drug: Skin antisepsis with chlorhexidine — Chlorhexidine swabs will be used to antiseptically clean the skin, then cultures of the skin and femoral nerve block catheters will be analyzed via standard microbiological techniques
  Other Names: Chlora-prep: 2% w/v chlorhexidine and 70% v/v isopropyl alcohol
  Arms: Chlorhexidine
Drug: povidone-iodine — Povidone-iodine swabs will be used to antiseptically clean the skin; then cultures of the skin and femoral nerve catheters will be performed by standard microbiologic techniques
  Other Names: Povidone-Iodine, USP 10% topical solution
  Arms: Povidone-iodine

SUMMARY:
Continuous femoral nerve block (CFNB) techniques continue to be increasingly used in the management of postoperative pain after total knee arthroplasty. Although the risk of full blown infection with CFNB has been poorly defined, the rate of catheter colonization after antisepsis with povidone-iodine has been demonstrated to be high (Cuivillion et al. showed the rate of colonization to be 57% after 48 hours). Recently, several anecdotal case reports have demonstrated severe infectious complications including psoas abscess and necrotizing fasciitis associated with continuous nerve block techniques. As the use of CFNB techniques increase in popularity, infectious complications will undoubtedly become more common.

The American Society of Regional Anesthesia and Pain Medicine recommends the routine use of antiseptic solutions with an alcohol base for skin disinfection before peripheral regional techniques due to their penetration of the stratum corneum and their rapid and prolonged effect. Chlorhexidine(chloraprep) has been proven to be better than povidone iodine solution for skin preparation before epidural catheter and intravascular device insertion (Kinirons et al., Ostrander et al., Mimoz et al.,). The goal of this prospective trial therefore is to determine if an alcoholic solution of 0.5% chlorhexidine is more effective than an aqueous solution of 10% povidone-iodine in reducing catheter colonization and reducing skin flora associated with short term ( 48 hours) postoperative continuous femoral nerve catheter placement. The investigators will also compare the ability of chloraprep and betadine disinfection at the time of catheter placement to prevent bacterial contamination of the continuous femoral catheter.

DETAILED DESCRIPTION:
After antisepsis four different cultures will be analyzed:

1. The femoral nerve catheter will be removed after 48 hours and a culture of the distal tip of the femoral nerve catheter will be performed between the 2 arms.
2. immediately before skin antisepsis, a culture of the the skin will be performed to identify baseline skin flora.
3. immediately after antisepsis with both betadine and chlorhexidine, a culture of the skin will be performed to assess antiseptic efficacy.
4. just prior to removal of the femoral nerve catheter, a culture of the skin/catheter interface will be performed between the 2 arms.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3,
* Undergoing primary total knee arthroplasty.

Exclusion Criteria:

* Hypersensitivity/allergy to antiseptics,
* Recent opioid/alcohol abuse,
* Presence of contraindications to regional anesthesia,
* Coagulation disorder,
* Diabetic/femoral neuropathy,
* Prior surgery to inguinal area,
* Patient refusal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Presence or absence of bacterial colonization of the distal femoral catheter tip 48 hours after antiseptic application | July 2013

SECONDARY OUTCOMES:
Incidences of bacterial colonization of skin before/after skin antisepsis and skin/catheter interface | July 2013

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Marino, M.D., Principal Investigator — Franklin Hospital
Locations (2):
- United States (2):
  - Syosset Hospital, Syosset, New York
  - Franklin Hospital, Valley Stream, New York